CLINICAL TRIAL: NCT01865929
Title: Benign Hysterectomy; a Randomized Controlled Trial Comparing Robotic Hysterectomy With Vaginal Hysterectomy and Traditional Laparoscopic Hysterectomy
Brief Title: Minimally Invasive Benign Hysterectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LundKK
Record Dates: First submitted 2013-04-08; First posted 2013-05-31 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-02

CONDITIONS: Menorrhagia; Metrorrhagia; Uterine Fibroids; Cervical Dysplasia
MeSH Terms: conditions — Menorrhagia; Metrorrhagia; Leiomyoma; Uterine Cervical Dysplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic hysterectomy (Active Comparator): Minimally invasive hysterectomy by robotic surgery
  Interventions: Procedure: Vaginal or laparoscopic hysterectomy
- Vaginal or laparoscopic hysterectomy (Active Comparator): Minimal invasive hysterectomy by vaginal or traditional laparoscopic surgery.
  Interventions: Device: Robotic hysterectomy

INTERVENTIONS:
Device: Robotic hysterectomy — Minimally invasive hysterectomy for benign disorders. Comparing robotic hysterectomy with vaginal hysterectomy and traditional laparoscopic hysterectomy
  Other Names: da Vinci Surgical system, Intuitive Surgical Inc, CA, USA
  Arms: Vaginal or laparoscopic hysterectomy
Procedure: Vaginal or laparoscopic hysterectomy — Benign hysterectomy performed by traditional minimal invasive procedures.
  Arms: Robotic hysterectomy

SUMMARY:
A randomised controlled trial comparing hysterectomy by minimally invasive surgical methods; robotic hysterectomy versus vaginal hysterectomy or traditional laparoscopic hysterectomy; outcome and cost analyses.

DETAILED DESCRIPTION:
Laparoscopic surgery is advantageous compared to open surgery in terms of patient morbidity, shorter hospitalization and a more rapid return to daily activities. Robot-assisted laparoscopic surgery have facilitated a higher proportion of minimally invasive surgery first and foremost within gynecologic oncology.It is not clear whether or not this is true for less advanced surgery where a vaginal approach or a traditional laparoscopic approach is possible.

Robot-assisted surgery is associated with additional cost due to investment and more expensive surgical equipment. The study is performed to investigate whether or not performing hysterectomy for benign conditions with robotic surgery will be advantageous in terms of shorter operating time, less complications, less conversions to open surgery, and shorter hospital stay in comparison to other minimally invasive procedures such as vaginal hysterectomy and traditional laparoscopic hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* indication for hysterectomy for benign disease or prophylactic surgery due to hereditary cancer
* size of uterus and vagina allows for retrieval by the vaginal route
* maximum uterine size equivalent to 16 weeks of pregnancy
* informed consent

Exclusion Criteria:

* malignant disease
* known extensive intra-abdominal adhesions
* anaesthesiological contraindications to laparoscopic surgery
* women with pacemaker or other implants where electrosurgery is to be avoided
* immunoincompetent women
* simultaneous need for prolapse surgery
* women with known defects of the hemostasis
* allergies towards metronidazole and doxycycline
* inability to understand patient information

Min Age: 25 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2010-01; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Cost of surgery | 4 months
  The cost of surgery includes the actual surgery (anaesthesia, OR-nurse, circulating nurse, doctors and use of the OR) as well as the length of the inpatient stay. The cost for conversions to open surgery, reoperations, readmissions, and any additional cost associated with additional procedures or medical interventions such as radiological examinations and blood transfusions. Based on the estimated cost of surgical material, use of the operating room and cost of anaesthesia each benign hysterectomy performed with robotic surgery would need to be 50 minutes shorter than other minimal invasive procedures to compensate for the additional cost.

SECONDARY OUTCOMES:
Patient outcome | 4 months
  The number of patients in whom an intraoperative or postoperative complication occurs as well as the seriousness of the complication which occurs and what this entails for the patient in question. This includes conversions to open surgery as well as the need for reoperation and readmission.

OTHER OUTCOMES:
Social cost | 4 months
  The length of postoperative sick leave and reasons for extending sick leave and cost thereof.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Persson, MD, PhD, Study Director — Department of Obstetrics and Gynecology, Skane University Hospital, Lund
Locations (1):
- Department of Obstetrics and Gynecology, Skane University Hospital, Lund, Sweden